CLINICAL TRIAL: NCT02909985
Title: Visual Activity Evoked by Infrared in Humans After Dark Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Olivia Hopkins, Assistant Professor-Clinical Educator, University of New Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CTSC0004-6
Record Dates: First submitted 2016-05-06; First posted 2016-09-21 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Age Related Macular Degeneration; Retinitis Pigmentosa; Congenital Stationary Night Blindness; Colorblindness
Keywords: Infrared; Dark Adaptation; Vision; Scotopic Threshold Response; Transient Receptor Potential (TRP) Channels; Human
MeSH Terms: conditions — Macular Degeneration; Retinitis Pigmentosa; Night blindness, congenital stationary; Color Vision Defects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual response to IR in healthy eyes (Experimental): 15 healthy participants will describe IR light passing through narrow bandpass filters over a broad-spectrum light source.
  As intensity increases from 0 to 12 V, participants will say if/when they see a visual response to infrared light from a broadband Tungsten halogen light with narrow bandpass filters ranging from 850 nm to 1400 nm. At the end of three trials per filter, the intensity will be turned up to 12 V, and participants will describe the color they see.
  Interventions: Other: Tungsten halogen light with narrow bandpass filters
- Visual response to IR in colorblind eyes (Experimental): 6 colorblind participants will describe IR light passing through narrow bandpass filters over a broad-spectrum light source.
  As intensity increases from 0 to 12 V, participants will say if/when they see a visual response to infrared light from a broadband Tungsten halogen light with narrow bandpass filters ranging from 850 nm to 1400 nm. At the end of three trials per filter, the intensity will be turned up to 12 V, and participants will describe the color they see.
  Interventions: Other: Tungsten halogen light with narrow bandpass filters

INTERVENTIONS:
Other: Tungsten halogen light with narrow bandpass filters — As intensity in increased from 0 to 12 V, participants will say if/when they see a visual response to infrared light from a broad band tungsten halogen light source that passes through narrow bandpass filters ranging from 850 nm to 1400 nm. At the end of three trials per filter, the intensity will be turned up to 12 V, and participants will describe the color they see.

SUMMARY:
This pilot study will evaluate the visual response to infrared (IR) in humans after dark adaptation. The investigators plan to determine which wavelength and intensity the human eye is most sensitive to in healthy and color-blind participants by using a broad spectrum light source and wavelength-specific IR bandpass filters.

The long-term goal of this research is to better understand the role that IR plays in visual function, and whether this can be manipulated to allow for vision in certain retinal pathologies that result from loss of photoreceptor cells. The investigators central objective is to test the electrophysiologic response to IR in the dark-adapted retinal and visual pathways. The investigator's central hypothesis is that IR evokes a visual response in humans after dark adaptation, and the characteristics of this response suggest transient receptor potential (TRP) channel involvement. The investigators rationale is that a better understanding of how IR impacts vision may allow for an alternative mechanism for vision in a number of diseases that cause blindness from the degradation or loss of function of photoreceptor cells. The investigators will test the investigator's hypothesis with the following Aims:

Aim 1:

Arm 1: To determine the optimal IR wavelength for visual perception in dark-adapted human participants. The investigators hypothesize that the healthy human eye will detect IR irradiation, with a maximum sensitivity at a specific wavelength. Using a broad-spectrum light source with wavelength-specific bandpass filters, the spectral range of visual perception to IR will be evaluated.

Arm 2: To determine the optimal IR wavelength for visual perception in dark-adapted human participants who are colorblind. The investigators hypothesize that the colorblind human eye will detect IR irradiation, with a maximum sensitivity at a specific wavelength. Using a broad-spectrum light source with wavelength-specific bandpass filters, the spectral range of visual perception to IR will be evaluated.

DETAILED DESCRIPTION:
BACKGROUND: Visual impairment affects 285 million people worldwide. The prevalence of visual impairment in the US is expected to rise from 3.3 million in 2000 to 5.5 million in 2020. This will exacerbate the current economic burden of vision loss, which is already $38.2 billion per year in direct and indirect costs. The leading cause of blindness in high-income countries is due to age-related macular degeneration (AMD), a disease that leads to gradual loss of the photoreceptor cell layer. An estimated 1.75 million people have AMD in the US and another 7.3 million are at risk. Importantly, despite the loss of photoreceptor cells in AMD, the other cellular layers in the retina remain largely intact.

The retina lines the back of the eye and is composed of structural layers. The outer nuclear layer contains photoreceptors called rods and cones. The inner nuclear layer includes bipolar, horizontal, and amacrine cells. Most anteriorly, the ganglion cell layer has axons that exit the eye as the optic nerve. Visual image formation begins when a photon of light enters the eye, passes through all retinal layers, and is absorbed by the photoreceptor cells. These cells transduce the photon of light into an electrochemical signal, which is communicated to bipolar cells, followed by the ganglion cells. Here, an action potential is generated and propagated via the optic nerve to the area of the brain where vision perception occurs. When the eye is dark-adapted, the cells in this pathway are potentially more sensitive to other types of stimuli, such as IR. The investigators believe cation channels called TRP channels in ganglion cells are activated by IR in this dark-adapted state, creating the visual response to IR. Heat is a known activator of certain subtypes of these channels elsewhere in the body. TRP channels are also responsible for IR vision in pit vipers and vampire bats.

Palczewska et al. reported that visual perception to IR occurred through a process of direct two-photon isomerization of visual pigments. However, other evidence suggests IR perception can occur through single IR photon absorption. Studies that use IR to test the functionality of implanted visual prosthesis have noted a greater response to IR in the non-implanted eye when compared to the implanted eye on both VEP tests and ERG. On ERG, a specialized response specific to IR was found called the scotopic threshold response (STR). This response occurs under dark-adapted conditions and correlates with a response at the ganglion cell layer. Direct IR activation of TRP channels on ganglion cells could initiate a visual response. Based on these findings, the investigators hypothesize the human response to IR under dark adaptation occurs at the level of the ganglion cells through heat-activated TRP channels.

RESEARCH DESIGN AIM1: To determine the optimal IR wavelength for human visual perception while dark-adapted in the healthy human eye.

Introduction for Aim 1: The objective of this aim is to determine the optimal wavelength of IR to which the human eye is sensitive. To obtain this objective, the investigators will test the working hypothesis that the healthy human eye, and those with colorblindness, will detect a range of IR wavelengths, with a preference for a specific wavelength. The investigators will test the working hypothesis using a broad-spectrum light source with wavelength-specific bandpass filters in the IR range. The investigators' rationale for this aim is that understanding the optimal IR wavelength of the human eye will aid in future investigations when testing the visual response to IR using diagnostic equipment. This is important because it could impact the way other ophthalmologic modalities use IR to diagnose and treat visual pathologies.

Research Design for Aim 1: A total of healthy 21 participants (15 with normal vision and 6 with colorblindness) aged 18 and older will be recruited using the University of New Mexico (UNM) Clinical and Translational Science Center (CTSC) Clinical Research Volunteer Registry HRRC-06412. Informed consent, participant demographics, past medial and visual history, and a general eye exam will be obtained using the CTSC research coordinator. Each participant will be placed in a dark room for an hour to allow for optimal dark adaptation of the eye. The investigators will use a broad-spectrum light source with wavelength-specific bandpass filters of different IR wavelengths. A total of 12 filters will be used ranging from 850 nm to 1400nm. Intensity curves will be built for each wavelength, by slowly turning up the power until the participant indicates a visual response to the stimulus.

Data Analysis for Aim 1: Data will be analyzed by the investigators. Descriptive statistics will be used to evaluate demographics, general and visual health information, and reported optimal wavelengths. The investigators' analysis will compare differences among responses for each wavelength. To the investigators' knowledge, there have been no studies evaluating which IR wavelength is optimal for human visual perception, thus the investigators assume a low effect size of 10%, which would produce an 82% chance of at least two out of 30 healthy participants giving a preferred response to a specific wavelength. The investigators will describe the estimated effect sizes in response to the findings.

Expected Outcomes for Aim 1: The investigators expect the human eye to perceive a range of IR wavelengths, but have a specific wavelength optimal in terms of brightness.

Potential Problems & Alternative Strategies for Aim 1: To prevent sampling bias, the investigators plan to obtain a representative sample from New Mexico; however, participants may be younger and more educated than the general population. The confounding bias of light pollution may occur, which would prevent dark adaptation and decrease the IR sensitivity. A photometer will assess the room for background photons.

ELIGIBILITY:
Inclusion Criteria:

* Normal Vision
* Colorblindness
* Age related macular degeneration
* Congenital Stationary Night Blindness

Exclusion Criteria:

* Diabetes
* Heart disease
* History of eye injury
* History of eye trauma
* History of eye disease except for those specified in the inclusion criteria
* Pregnant women will also be excluded from Aim 2 and 3
* Persons with allergies to adhesives will be excluded from Aim 2 and 3
* Contact dermatitis
* Documented adverse reaction to dilating drops
* Documented adverse reaction to topical anesthetics
* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Olivia Hopkins, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittenborn JS, Zhang X, Feagan CW, Crouse WL, Shrestha S, Kemper AR, Hoerger TJ, Saaddine JB; Vision Cost-Effectiveness Study Group. The economic burden of vision loss and eye disorders among the United States population younger than 40 years. Ophthalmology. 2013 Sep;120(9):1728-35. doi: 10.1016/j.ophtha.2013.01.068. Epub 2013 Apr 28. PMID 23631946
- [Background] Pascolini D, Mariotti SP. Global estimates of visual impairment: 2010. Br J Ophthalmol. 2012 May;96(5):614-8. doi: 10.1136/bjophthalmol-2011-300539. Epub 2011 Dec 1. PMID 22133988
- [Background] Stockman A, Sharpe LT, Fach C. The spectral sensitivity of the human short-wavelength sensitive cones derived from thresholds and color matches. Vision Res. 1999 Aug;39(17):2901-27. doi: 10.1016/s0042-6989(98)00225-9. PMID 10492818
- [Background] Friedman DS, O'Colmain BJ, Munoz B, Tomany SC, McCarty C, de Jong PT, Nemesure B, Mitchell P, Kempen J; Eye Diseases Prevalence Research Group. Prevalence of age-related macular degeneration in the United States. Arch Ophthalmol. 2004 Apr;122(4):564-72. doi: 10.1001/archopht.122.4.564. PMID 15078675
- [Background] White JP, Urban L, Nagy I. TRPV1 function in health and disease. Curr Pharm Biotechnol. 2011 Jan 1;12(1):130-44. doi: 10.2174/138920111793937844. PMID 20932253
- [Background] Numazaki M, Tominaga M. Nociception and TRP Channels. Curr Drug Targets CNS Neurol Disord. 2004 Dec;3(6):479-85. doi: 10.2174/1568007043336789. PMID 15578965
- [Background] Gracheva EO, Ingolia NT, Kelly YM, Cordero-Morales JF, Hollopeter G, Chesler AT, Sanchez EE, Perez JC, Weissman JS, Julius D. Molecular basis of infrared detection by snakes. Nature. 2010 Apr 15;464(7291):1006-11. doi: 10.1038/nature08943. Epub 2010 Mar 14. PMID 20228791
- [Background] Gekeler F, Shinoda K, Blatsios G, Werner A, Zrenner E. Scotopic threshold responses to infrared irradiation in cats. Vision Res. 2006 Feb;46(3):357-64. doi: 10.1016/j.visres.2005.06.023. Epub 2005 Aug 2. PMID 16081127
- [Background] Pardue MT, Ball SL, Hetling JR, Chow VY, Chow AY, Peachey NS. Visual evoked potentials to infrared stimulation in normal cats and rats. Doc Ophthalmol. 2001 Sep;103(2):155-62. doi: 10.1023/a:1012202410144. PMID 11720256
- [Background] Chow AY, Pardue MT, Chow VY, Peyman GA, Liang C, Perlman JI, Peachey NS. Implantation of silicon chip microphotodiode arrays into the cat subretinal space. IEEE Trans Neural Syst Rehabil Eng. 2001 Mar;9(1):86-95. doi: 10.1109/7333.918281. PMID 11482368
- [Background] Sieving PA, Frishman LJ, Steinberg RH. Scotopic threshold response of proximal retina in cat. J Neurophysiol. 1986 Oct;56(4):1049-61. doi: 10.1152/jn.1986.56.4.1049. PMID 3783228
- [Background] Wakabayashi K, Gieser J, Sieving PA. Aspartate separation of the scotopic threshold response (STR) from the photoreceptor a-wave of the cat and monkey ERG. Invest Ophthalmol Vis Sci. 1988 Nov;29(11):1615-22. PMID 3182196
- [Background] Kolb H. Simple Anatomy of the Retina. 2005 May 1 [updated 2012 Jan 31]. In: Kolb H, Fernandez E, Jones B, Nelson R, editors. Webvision: The Organization of the Retina and Visual System [Internet]. Salt Lake City (UT): University of Utah Health Sciences Center; 1995-. Available from http://www.ncbi.nlm.nih.gov/books/NBK11533/ PMID 21413391
- [Background] Palczewska G, Vinberg F, Stremplewski P, Bircher MP, Salom D, Komar K, Zhang J, Cascella M, Wojtkowski M, Kefalov VJ, Palczewski K. Human infrared vision is triggered by two-photon chromophore isomerization. Proc Natl Acad Sci U S A. 2014 Dec 16;111(50):E5445-54. doi: 10.1073/pnas.1410162111. Epub 2014 Dec 1. PMID 25453064
- See also: ARVO Meeting Abstract — http://iovs.arvojournals.org/article.aspx?articleid=2409738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult participants with normal vision or who are colorblind were recruited using the University of New Mexico CTSC Clinical Research Volunteer Registry (HRRC 06-412), a Craigslist advertisement, and word of mouth.
Groups:
- Visual Response to IR: 1. 15 healthy participants described IR light passing through narrow bandpass filters over a broad spectrum light source
  2. 6 colorblind participants described IR light passing through narrow bandpass filters over a broad spectrum light source
  All participants signed informed consent, demographics, general and visual health information, and a Snellen eye exam was collected. An Ishihara Plate Test and modified Farnsworth D-15 test were obtained for those with color blindness.
  For both groups, as the intensity was increased from 0 to 12 V, participants said if/when they saw a visual response to infrared light from a broadband Tungsten halogen light with narrow bandpass filters ranging from 850 nm to 1400 nm. At the end of three trials per filter, the intensity was turned up to 12 V, and participants described the color they saw.
Period: Overall Study
Arm/Group | Visual Response to IR
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Visual Response to IR in Colorvision Eyes: The goal of this aim is to determine which wavelength and intensity of IR the human eye with normal color vision is most sensitive to. This arm includes those with normal color vision who will be exposed to a range of IR wavelengths using a broad-spectrum light source with wavelength-specific bandpass filters in the IR range. Participants will give verbal feedback on when they can see the stimulus over three trials at each wavelength, and then describe the color they see when the light is set at 12 V.
- Visual Response to IR in Colorblind Eyes: The goal of this aim is to determine which wavelength and intensity of IR the human eye with colorblindness is most sensitive to. This arm includes those with colorblind vision who will be exposed to a range of IR wavelengths using a broad-spectrum light source with wavelength-specific bandpass filters in the IR range. Participants will give verbal feedback on when they can see the stimulus over three trials at each wavelength, and then describe the color they see when the light is set at 12 V.
- Total: Total of all reporting groups
Arm/Group | Visual Response to IR in Colorvision Eyes | Visual Response to IR in Colorblind Eyes | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 5 | 20
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 37.6 [22 to 58] | 45.7 [27 to 71] | 40 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 9 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 12 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 13 | 5 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Visual Perception to Infrared: Mean Minimal Intensity (uW) at Which Participants Could See IR Between 900 - 1400 nm.
Description: We measured the minimum threshold intensities (uW) via subjective perception of near IR light (900 - 1400 nm) in 50 nm intervals. After 30 minutes of dark adaptation and over three trials, participants verbalized by saying 'yes' to the minimal intensity they could see the IR stimulus as the power source for the light was slowly increased from 0V to 12 V. The voltage was averaged for the three trials at each wavelength. Analysis of variance was used to evaluate the effect of the wavelength on the threshold intensity. This was done for two groups/arms, one with normal color vision and one with colorblind vision.
Time Frame: after 30 minutes of dark adaptation, up to 2 hours
Population: Adults with normal color vision and colorblind vision were evaluated for the minimal threshold intensity (uW) at which they could subjectively perceive IR as the light was slowly increased from 0-12 V. The average of three trials per IR wavelength was obtained.
Measure: Mean (Standard Deviation); unit: uW
Groups:
- Normal Color Vision; Colorblind Vision: Average of minimal intensity at which participants would see the IR stimulus for three trials at each wavelength. Analysis of variance was used to evaluate the effect of the wavelength on the threshold intensity.
Arm/Group | Normal Color Vision | Colorblind Vision
Number analyzed (Participants) | 15 | 6
uW
  850 nm | 0.671770454 (0.099031306) | 0.809204 (0.141801)
  900 nm | 0.205456012 (0.037481007) | 0.222247 (0.042895)
  950 nm | 0.281608408 (0.070729646) | 0.545299 (0.571049)
  1000 nm | 1.144748348 (0.607965504) | 1.056031 (0.792399)
  1050 nm | 1.272084129 (0.672594905) | 1.397371 (0.90500)
  1100 nm | 0.258018884 (0.089276004) | 0.367814 (0.205764)
  1150 nm | 1.353030502 (0.911531487) | 2.144498 (1.049761)
  1200 nm | 0.345439815 (0.143985558) | 0.422416 (0.119660)
  1250 nm | 0.341422349 (0.194358383) | 0.505195 (0.229724)
  1300 nm | 0.153133406 (0.097493319) | 0.198776 (0.095276)
  1350 nm | 0.119277641 (0.0881392) | 0.182666 (0.067348)
  1400 nm | 0.419039248 (0.158978102) | 0.601534 (0.184694)
Statistical Analysis 1: Comparison: Normal Color Vision; Test type: Superiority; p < 0.0001, ANOVA; (9, 129); F = 23.68
Statistical Analysis 2: Comparison: Colorblind Vision; Test type: Superiority; p < 0.0001, ANOVA; (11, 52); F = 9.4394

2. Secondary Outcome: Description of Color
Description: A subjective description of color was given by each participant for each wavelength between 850 - 1400nm while at 12V.
Time Frame: after 30 minutes of dark adaptation, up to 2 hours
Population: Adult participants who have normal color vision and those who are colorblind will be dark adapted for 30 minutes and then complete outcome measure 1 followed by outcome measure 2, in which the light source will be increased to a maximum of 12 V, and the participant will give a subjective description of color for each wavelength between 850 - 1400 nm in 50nm increments.
  Note* Unable to add color chart results reported as 'color' to outcome measure data table.
Measure: Count of Participants; unit: Participants
Groups:
- Visual Response to IR in Colorvision Eyes: 15 participants with normal color vision will give a subjective description of color for each wavelength between 850 - 1400nm while the light is at a maximum of 12V.
- Visual Response to IR in Colorblind Eyes: 6 colorblind participants will describe IR light passing through narrow bandpass filters over a broad-spectrum light source.
  6 participants with colorblind vision will give a subjective description of color for each wavelength between 850 - 1400nm while the light is at a maximum of 12V.
Arm/Group | Visual Response to IR in Colorvision Eyes | Visual Response to IR in Colorblind Eyes
Number analyzed (Participants) | 15 | 6
Participants
  Color perception at 850 λ: Red | 12 | 4
  Color perception at 850 λ: Dark Red | 3 | 0
  Color perception at 850 λ: Orange | 0 | 1
  Color perception at 850 λ: Yellow | 0 | 0
  Color perception at 850 λ: Light brown | 0 | 0
  Color perception at 850 λ: Light blue | 0 | 0
  Color perception at 850 λ: Blue | 0 | 0
  Color perception at 850 λ: Light Purple | 0 | 0
  Color perception at 850 λ: White | 0 | 0
  Color perception at 850 λ: Grey | 0 | 0
  Color perception at 850 λ: Teal Green | 0 | 0
  Color perception at 850 λ: Green | 0 | 1
  Color perception at 850 λ: Light Green | 0 | 0
  Color perception at 850 λ: Black (no color) | 0 | 0
  Color perception at 850 λ: Pink | 0 | 0
  Color perception at 900 λ: Red | 4 | 1
  Color perception at 900 λ: Dark Red | 1 | 0
  Color perception at 900 λ: Orange | 7 | 2
  Color perception at 900 λ: Yellow | 0 | 0
  Color perception at 900 λ: Light brown | 0 | 0
  Color perception at 900 λ: Light blue | 0 | 0
  Color perception at 900 λ: Blue | 0 | 0
  Color perception at 900 λ: Light Purple | 0 | 0
  Color perception at 900 λ: White | 0 | 0
  Color perception at 900 λ: Grey | 0 | 0
  Color perception at 900 λ: Teal Green | 0 | 1
  Color perception at 900 λ: Green | 0 | 1
  Color perception at 900 λ: Light Green | 0 | 1
  Color perception at 900 λ: Black (no color) | 1 | 0
  Color perception at 900 λ: Pink | 2 | 0
  Color perception at 950 λ: Red | 0 | 1
  Color perception at 950 λ: Dark Red | 1 | 0
  Color perception at 950 λ: Orange | 4 | 0
  Color perception at 950 λ: Yellow | 2 | 2
  Color perception at 950 λ: Light brown | 5 | 0
  Color perception at 950 λ: Light blue | 0 | 0
  Color perception at 950 λ: Blue | 0 | 0
  Color perception at 950 λ: Light Purple | 1 | 0
  Color perception at 950 λ: White | 1 | 0
  Color perception at 950 λ: Grey | 0 | 1
  Color perception at 950 λ: Teal Green | 0 | 0
  Color perception at 950 λ: Green | 0 | 0
  Color perception at 950 λ: Light Green | 0 | 1
  Color perception at 950 λ: Black (no color) | 0 | 0
  Color perception at 950 λ: Pink | 1 | 1
  Color perception at 1000 λ: Red | 1 | 0
  Color perception at 1000 λ: Dark Red | 0 | 0
  Color perception at 1000 λ: Orange | 1 | 0
  Color perception at 1000 λ: Yellow | 0 | 0
  Color perception at 1000 λ: Light brown | 0 | 0
  Color perception at 1000 λ: Light blue | 1 | 0
  Color perception at 1000 λ: Blue | 0 | 0
  Color perception at 1000 λ: Light Purple | 0 | 0
  Color perception at 1000 λ: White | 1 | 1
  Color perception at 1000 λ: Grey | 0 | 0
  Color perception at 1000 λ: Teal Green | 1 | 0
  Color perception at 1000 λ: Green | 0 | 0
  Color perception at 1000 λ: Light Green | 0 | 0
  Color perception at 1000 λ: Black (no color) | 10 | 5
  Color perception at 1000 λ: Pink | 0 | 0
  Color perception at 1050 λ: Red | 0 | 0
  Color perception at 1050 λ: Dark Red | 0 | 0
  Color perception at 1050 λ: Orange | 0 | 0
  Color perception at 1050 λ: Yellow | 0 | 0
  Color perception at 1050 λ: Light brown | 0 | 0
  Color perception at 1050 λ: Light blue | 2 | 0
  Color perception at 1050 λ: Blue | 0 | 0
  Color perception at 1050 λ: Light Purple | 0 | 0
  Color perception at 1050 λ: White | 3 | 0
  Color perception at 1050 λ: Grey | 0 | 1
  Color perception at 1050 λ: Teal Green | 2 | 0
  Color perception at 1050 λ: Green | 0 | 0
  Color perception at 1050 λ: Light Green | 0 | 0
  Color perception at 1050 λ: Black (no color) | 8 | 5
  Color perception at 1050 λ: Pink | 0 | 0
  Color perception at 1100 λ: Red | 0 | 0
  Color perception at 1100 λ: Dark Red | 0 | 0
  Color perception at 1100 λ: Orange | 2 | 1
  Color perception at 1100 λ: Yellow | 5 | 1
  Color perception at 1100 λ: Light brown | 0 | 0
  Color perception at 1100 λ: Light blue | 0 | 0
  Color perception at 1100 λ: Blue | 0 | 0
  Color perception at 1100 λ: Light Purple | 1 | 0
  Color perception at 1100 λ: White | 3 | 0
  Color perception at 1100 λ: Grey | 2 | 1
  Color perception at 1100 λ: Teal Green | 0 | 0
  Color perception at 1100 λ: Green | 0 | 1
  Color perception at 1100 λ: Light Green | 0 | 1
  Color perception at 1100 λ: Black (no color) | 1 | 0
  Color perception at 1100 λ: Pink | 1 | 1
  Color perception at 1150 λ: Red | 1 | 0
  Color perception at 1150 λ: Dark Red | 0 | 0
  Color perception at 1150 λ: Orange | 0 | 1
  Color perception at 1150 λ: Yellow | 0 | 0
  Color perception at 1150 λ: Light brown | 1 | 0
  Color perception at 1150 λ: Light blue | 1 | 0
  Color perception at 1150 λ: Blue | 1 | 0
  Color perception at 1150 λ: Light Purple | 0 | 1
  Color perception at 1150 λ: White | 6 | 2
  Color perception at 1150 λ: Grey | 2 | 1
  Color perception at 1150 λ: Teal Green | 1 | 0
  Color perception at 1150 λ: Green | 0 | 0
  Color perception at 1150 λ: Light Green | 0 | 1
  Color perception at 1150 λ: Black (no color) | 2 | 0
  Color perception at 1150 λ: Pink | 0 | 0
  Color perception at 1200 λ: Red | 1 | 1
  Color perception at 1200 λ: Dark Red | 4 | 0
  Color perception at 1200 λ: Orange | 5 | 1
  Color perception at 1200 λ: Yellow | 1 | 1
  Color perception at 1200 λ: Light brown | 1 | 0
  Color perception at 1200 λ: Light blue | 0 | 0
  Color perception at 1200 λ: Blue | 1 | 0
  Color perception at 1200 λ: Light Purple | 0 | 0
  Color perception at 1200 λ: White | 1 | 0
  Color perception at 1200 λ: Grey | 0 | 1
  Color perception at 1200 λ: Teal Green | 0 | 1
  Color perception at 1200 λ: Green | 0 | 0
  Color perception at 1200 λ: Light Green | 0 | 1
  Color perception at 1200 λ: Black (no color) | 1 | 0
  Color perception at 1200 λ: Pink | 0 | 0
  Color perception at 1250 λ: Red | 1 | 0
  Color perception at 1250 λ: Dark Red | 4 | 0
  Color perception at 1250 λ: Orange | 6 | 1
  Color perception at 1250 λ: Yellow | 1 | 1
  Color perception at 1250 λ: Light brown | 1 | 0
  Color perception at 1250 λ: Light blue | 0 | 0
  Color perception at 1250 λ: Blue | 0 | 1
  Color perception at 1250 λ: Light Purple | 1 | 0
  Color perception at 1250 λ: White | 0 | 0
  Color perception at 1250 λ: Grey | 0 | 1
  Color perception at 1250 λ: Teal Green | 0 | 0
  Color perception at 1250 λ: Green | 0 | 1
  Color perception at 1250 λ: Light Green | 0 | 1
  Color perception at 1250 λ: Black (no color) | 1 | 0
  Color perception at 1250 λ: Pink | 0 | 0
  Color perception at 1300 λ: Red | 11 | 1
  Color perception at 1300 λ: Dark Red | 1 | 0
  Color perception at 1300 λ: Orange | 1 | 2
  Color perception at 1300 λ: Yellow | 0 | 2
  Color perception at 1300 λ: Light brown | 0 | 0
  Color perception at 1300 λ: Light blue | 0 | 0
  Color perception at 1300 λ: Blue | 0 | 0
  Color perception at 1300 λ: Light Purple | 0 | 0
  Color perception at 1300 λ: White | 0 | 0
  Color perception at 1300 λ: Grey | 0 | 0
  Color perception at 1300 λ: Teal Green | 0 | 0
  Color perception at 1300 λ: Green | 0 | 1
  Color perception at 1300 λ: Light Green | 0 | 0
  Color perception at 1300 λ: Black (no color) | 1 | 0
  Color perception at 1300 λ: Pink | 1 | 0
  Color perception at 1350 λ: Red | 10 | 2
  Color perception at 1350 λ: Dark Red | 3 | 0
  Color perception at 1350 λ: Orange | 0 | 1
  Color perception at 1350 λ: Yellow | 0 | 1
  Color perception at 1350 λ: Light brown | 0 | 0
  Color perception at 1350 λ: Light blue | 0 | 0
  Color perception at 1350 λ: Blue | 0 | 0
  Color perception at 1350 λ: Light Purple | 0 | 0
  Color perception at 1350 λ: White | 0 | 0
  Color perception at 1350 λ: Grey | 0 | 0
  Color perception at 1350 λ: Teal Green | 0 | 0
  Color perception at 1350 λ: Green | 0 | 2
  Color perception at 1350 λ: Light Green | 0 | 0
  Color perception at 1350 λ: Black (no color) | 1 | 0
  Color perception at 1350 λ: Pink | 1 | 0
  Color perception at 1400 λ: Red | 6 | 1
  Color perception at 1400 λ: Dark Red | 0 | 1
  Color perception at 1400 λ: Orange | 6 | 1
  Color perception at 1400 λ: Yellow | 1 | 0
  Color perception at 1400 λ: Light brown | 0 | 0
  Color perception at 1400 λ: Light blue | 0 | 0
  Color perception at 1400 λ: Blue | 0 | 0
  Color perception at 1400 λ: Light Purple | 0 | 0
  Color perception at 1400 λ: White | 0 | 0
  Color perception at 1400 λ: Grey | 0 | 1
  Color perception at 1400 λ: Teal Green | 0 | 0
  Color perception at 1400 λ: Green | 0 | 2
  Color perception at 1400 λ: Light Green | 0 | 0
  Color perception at 1400 λ: Black (no color) | 1 | 0
  Color perception at 1400 λ: Pink | 1 | 0

ADVERSE EVENTS:
Time Frame: The study started on 9/2015 and was completed on 8/2016, during which time the adverse event data was monitored. Each participant was assessed during their participation in the study for up to two hours.
Groups:
- Visual Response to IR: There were no adverse events to report in this study.
Arm/Group | Visual Response to IR
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
Color descriptions vary among individuals. Our sample size was too small to permit any assessment of gender bias.

We were unable to standardize color descriptions with a reference color chart, as it was important to maintain dark adaptation in our participants. A color chart likely would have made this data more meaningful in understanding the colors reported and perceived by these participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes